CLINICAL TRIAL: NCT07404163
Title: The Effect of a Walkway Used in Postoperative Mobilization on Children's Pain, Fear, and Time to Initiate Mobilization
Brief Title: Walkway Used in Postoperative Mobilization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Esra AYDIN, MSc, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2026-04
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pain; Fear; Children; Surgery; Mobilization
Keywords: pain; Fear; Children; surgery; Mobilization
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walkway group (Experimental): In the experimental group, a washable/disinfectable mat with colorful figures and a target route will be placed in front of the children's beds. The child will be mobilized using this track in addition to standard parental support.
  Interventions: Other: Walkway
- no intervention (No Intervention): Control Group: Mobilization will be provided with parental support as part of the clinic's routine.

INTERVENTIONS:
Other: Walkway — In the experimental group, a washable/disinfectable mat with colorful figures and a target route will be placed in front of the children's beds.
  Arms: Walkway group

SUMMARY:
Introduction Surgical operations are increasing globally, with abdominal surgeries accounting for approximately 70% of these procedures. Despite the prevalence, postoperative complications occur in 30-60% of cases, leading to prolonged hospital stays, increased mortality, and higher healthcare costs. Early mobilization is a critical component of Enhanced Recovery After Surgery (ERAS) protocols, known to reduce surgical stress, muscle atrophy, and pulmonary complications. However, implementation in pediatric care is often limited, as children may perceive mobilization as a "task" rather than a part of healing.

Purpose The primary aim of this study is to investigate the effects of a low-cost, distraction-based Walkway (Mat Carpet) on pain levels, fear, and the time to initiate mobilization in children aged 4-10 who have undergone abdominal surgery.

DETAILED DESCRIPTION:
Early mobilization is defined as the patient's ability to stand up and walk as soon as possible after surgery or after illness, depending on the type of operation performed and the course of the disease. Early mobilization is considered and recommended as one of the factors that accelerate recovery. One study indicated that initiating movement and mobilization early reduced surgical stress, muscle atrophy, complications, hospital stay, and care costs. Other studies have also reported that early mobilization accelerates the functioning of the Gastrointestinal System (GIS), prevents thromboembolic complications, and speeds up recovery. To minimize complications after surgery and optimize the child's health, the Enhanced Recovery After Surgery (ERAS) protocol can be applied. These protocols, also known as "Fast-Track," were first implemented in 2001. Early mobilization is one of the most important components of the ERAS approach. According to the ERAS protocol, the patient needs to be mobilized for two hours on the day of surgery and for a total of six hours on subsequent days until discharge.

Although the benefits of early mobilization after surgery and its contribution to the recovery process are known, one study reported that early mobilization attempts were infrequent for patients after surgery (Rafeeqi and Pearson, 2021). Another study also indicated that patients need assistance with mobilization after surgical operations. At this point, nurses are key in initiating the early mobilization process to improve the quality of postoperative care. It is essential that early mobilization is initiated by the nurse, followed by encouraging the child to move independently. The surgical nurse should support the patient to achieve the highest possible level of independence and help improve their well-being.

Randomized controlled trials that comprehensively assess both physical performance and psychological comfort (pain and fear) simultaneously during mobilization in postoperative children are limited. This study is designed as a randomized controlled trial to prove the effectiveness of low-cost, easy-to-implement, and concrete play materials such as "Walking Tracks" (Mat Mats), which are distraction-based and suitable for children's developmental characteristics, in contrast to expensive and technology-based mobilization initiatives in the literature. It aims to fill the evidence gap that holistically evaluates both physical and psychological recovery. This study aims to improve both physical and psychological recovery in a holistic way by transforming mobilization in children from a "task" into a "game". The population of the study, which is planned as a randomized controlled trial, will consist of 74 children aged 4-10 years who underwent abdominal surgery in the Pediatric Surgery Department of Mersin University Hospital.

Methodology

Study Design: A randomized controlled experimental design will be employed.

Setting & Sample: The study will be conducted at Mersin University Hospital Pediatric Surgery Service. A total of 74 children (37 experiment, 37 control) will be recruited based on power analysis.

Randomization: Stratified block randomization will be used based on Surgical Technique (Open vs. Laparoscopic) and Developmental Stage (4-6 years vs. 7-10 years) to ensure group homogeneity.

Intervention: The experimental group will use a "Walkway" mat featuring colorful figures and a target route placed in front of their beds. The control group will receive standard parent-supported mobilization.

Data Collection Tools: * Introductory Information Form

Wong-Baker FACES Pain Rating Scale

Children's Fear Scale

Vital Signs Tracking Form

Procedure: A pilot study with 10 children will precede the main study. Mobilization for all participants will begin 30-60 minutes after a standard dose of analgesic (paracetamol) to ensure comfort. Pain and fear will be assessed by the child, parent, and nurse simultaneously before and after mobilization.

Statistical Analysis Data will be analyzed using SPSS, employing descriptive statistics, t-tests, or Mann-Whitney U tests for group comparisons. Consistency between child, parent, and nurse assessments will be measured using the Cohen's Kappa Test.

Expected Outcomes It is hypothesized that turning mobilization into a game via the walkway will significantly reduce the children's fear and pain levels while shortening the time to initiate the first step. This study aims to provide nursing evidence for holistic, low-cost, and developmentally appropriate pediatric postoperative care.

ELIGIBILITY:
Inclusion Criteria:

* Being between 4-10 years old
* Having undergone abdominal surgery
* Having undergone surgery under general anesthesia
* Having received analgesics (paracetamol) after surgery
* Having undergone initial mobilization after surgery
* Being a volunteer to participate in the study

Exclusion Criteria:

* Having undergone previous surgery
* A parent having undergone abdominal surgery
* The child having visual, hearing, or intellectual disabilities

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2026-02-04 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Wong Baker Pain Scale | 1 day
  Developed in 1981 by Donna Wong and Connie Morain Baker and revised in 1983, this scale is designed to assess children's pain levels. It includes six facial expressions scored from zero to ten.
Fear Scale | 1 day
  Developed by Thurillet et al. to assess children's fears based on self-reports from children aged 4-12 years. The Turkish validity and reliability study was conducted by Tavşan et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tazreean, R., Nelson, G., & Twomey, R. (2021). Early mobilization in enhanced recovery after surgery pathways: current evidence and recent advancements. Journal of Comparative Effectiveness Research, 11(2), 121-129.
- [Background] Wijk, L. (2022). Early mobilization and impact on recovery. In The ERAS® Society Handbook for Obstetrics & Gynecology (pp. 177-192). Academic Press.
- [Background] Townsend, C. M., Beauchamp, R. D., Evers, B. M., & Mattox, K. L. (2022). Sabiston textbook of surgery: The biological basis of modern surgical practice (21. baskı). Elsevier.
- [Background] Holcomb, G. W., Murphy, J. P., & St. Peter, S. D. (2020). Holcomb and Ashcraft's pediatric surgery (7. baskı). Elsevier.
- [Background] Kırtıl, İ., Kanan, N., & Karip, A. B. (2023). Effects of a mobilization program applied to bariatric surgery patients on preventing gastrointestinal complications: a quasi-experimental study. Obesity Surgery, 33(6), 1820-1830.
- [Background] Rafeeqi, T., & Pearson, E. G. (2021). Enhanced recovery after surgery in children. Translational gastroenterology and hepatology, 6, 46. https://doi.org/10.21037/tgh-20-188
- [Background] Akdağ, Y. M. (2019). Akut apendisit ameliyatı olan 6-12 yaş grubu çocukların postoperatif dönemde çevre oyunu ile mobilizasyonunun korku ve ağrı düzeyine etkisi (Yüksek lisans tezi). İstanbul Okan Üniversitesi.
- [Background] Daldaban, F. N. (2023). Erken mobilizasyon eğitiminin abdominal cerrahi sonrası hareketlilik, ağrı ve konfor üzerine etkisi (Yüksek lisans tezi). Doğu Akdeniz Üniversitesi.